CLINICAL TRIAL: NCT02895451
Title: Behavioral Interventions for Improvement of Adherence at Exercise-based Cardiac Rehabilitation (ECRA)
Acronym: ECRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Maria Bäck, PhD, RPT, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr: 2015/209-31
Record Dates: First submitted 2016-08-16; First posted 2016-09-09 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
Keywords: Exercise-based cardiac rehabilitation; Physical capacity; Adherence; Behavioral medicine
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended behavioral intervention (Experimental): Specific goal-setting, self-monitoring and feed-back
  Interventions: Behavioral: Extended behavioral intervention
- Usual care (No Intervention): Hospital-based or home-based aerobic exercise 3 times a week with a duration of 30-60 minutes and an intensity of 40-80 % of Vo2max and resistance exercise 2 times a week of 1-3 sets of 10-15 repetitions. The exercise period is 16 weeks.

INTERVENTIONS:
Behavioral: Extended behavioral intervention — The exercise goal is set in liaison between the patient and the physiotherapist, based on activities and target behaviors that the patient thinks is relevant and important. The patients are asked to self-monitor the defined exercise goal by completing an exercise diary. The exercise diary includes specification of the performed exercise dose (frequency, intensity and duration). The exercise diary is followed up by a physiotherapist every third week by a phone call or a personal meeting. Visual feed-back on the performed dose of exercise is given once by accelerometry. At end of intervention (16 weeks) the patient is offered a follow-up meeting with the physiotherapist to discuss a long-term exercise goal.
  Arms: Extended behavioral intervention

SUMMARY:
The purpose of this study is to investigate the effects of an extended behavioral intervention in exercise-based CR for improvement of physical capacity, adherence, psychological and physiological parameters, compared with usual care.

DETAILED DESCRIPTION:
Consecutive patients will be included at the coronary care unit (CCU), Linköping University Hospital, Sweden. Physiotherapists ask patients for informed consent at the CCU and book an appointment at the exercise-based CR 2-3 weeks after discharge for baseline tests. After baseline testing patients will be randomized to either extended intervention or routine care. Randomization will be stratified by submaximal exercise capacity. Patients randomized to the extended intervention group receive an additional appointment to a physiotherapist within a week. Thereafter patients in both groups start the exercise-based CR program, including aerobic exercise and resistance exercise, 3 times/week for 16 weeks, according to international guidelines for exercise-based CR.

The extended intervention is based on components from behavioral medicine including: specific goal-setting, self-monitoring and feed-back.

Changes in the endpoint variables will be measured from baseline to first (16 weeks at end of intervention) and second (12 months after index event) follow-up visits.

Sample size calculations are based on previous clinical data from a similar exercise-based CR setting (n=50) on differences in aerobic exercise capacity measured by submaximal exercise test (watts) before vs after finished exercise-based CR. With a power of 80% and a two-sided significance level of p<0.05 and least mean difference at 10 watts (SD 20 watts) and a calculated loss of follow-up of 20%, the estimated sample size is 160 patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary care event due to coronary artery disease and/or percutaneous coronary intervention (PCI) at the coronary care unit, Linköping University hospital
* Age <75 years

Exclusion Criteria:

* Serious physical or psychological disease interfering with participation in exercise-based CR
* Inability to understand the Swedish language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-12-15; Primary Completion 2019-04-15 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline aerobic exercise capacity (watts) at 4 months | 4 months
  The test is performed on a bicycle ergometer according to the WHO-protocol with an increased workload of 25W every 4.5 minutes.The exercise test is discontinued at Borg RPE 17 and/or dyspnea 7 at Borg´s CR-10 scale.

SECONDARY OUTCOMES:
Adherence to dose of exercise | 4 months
  accelerometer
Adherence to dose in exercise | 4 months
  exercise diary
Change from baseline unilateral isotonic shoulder flexion (repetitions) at 4 months | 4 months
  Muscle endurance test
Change from baseline unilateral isotonic heel lift (repetitions) at 4 months | 4 months
  Muscle endurance test
Change from baseline anxiety score at 4 months | 4 months
  Hospital Anxiety and Depression Scale (HADS)
Change from baseline depression score at 4 months | 4 months
  Hospital Anxiety and Depression Scale (HADS)
Change from baseline self-efficacy score at 4 months | 4 months
  Self Efficacy Exercise Scale (SEE-SV)
Change from baseline health-related quality of life score at 4 months | 4 months
  Short-Form-36 (SF-36)
Change from baseline health-related quality of life score at 4 months | 4 months
  EQ5D
Change from baseline level of physical activity at 4 months | 4 months
  Accelerometer
Change from baseline level of physical activity at 4 months | 4 months
  Bouchard questionnaire
Change from baseline aerobic exercise capacity (watts) at 12 months | 12 months
  Submaximal exercise test on bicycle ergometer
Adherence to dose of exercise | 12 months
  Accelerometer
Adherence to dose of exercise | 12 months
  Exercise diary
Change from baseline unilateral isotonic shoulder flexion (repetitions) at 12 months | 12 months
  Muscle endurance test
Change from baseline unilateral isotonic heel lift (repetitions) at 12 months | 12 months
  Muscle endurance test
Change from baseline anxiety score at 12 months | 12 months
  Hospital Anxiety and Depression Scale (HADS)
Change from baseline depression score at 12 months | 12 months
  Hospital Anxiety and Depression Scale (HADS)
Change from baseline self-efficacy score at 12 months | 12 months
  Self Efficacy Exercise Scale (SEE-SV)
Change from baseline health-related quality of life score at 12 months | 12 months
  Short-Form-36 (SF-36)
Change from baseline health-related quality of life score at 12 months | 2 months
  EQ5D
Change from baseline level of physical activity at 12 months | 12 months
  accelerometer
Change from baseline level of physical activity at 12 months | 12 months
  Bouchard questionnaire
Patient Enablement (score) | 12 months
  Patient Enablement Instrument (PEI)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bäck, PhD, Study Chair — Linkoeping University, Department of Medical and Health Sciences, Division of Physiotherapy
Locations (1):
- Linkoeping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borg S, Oberg B, Nilsson L, Alfredsson J, Soderlund A, Back M. Effectiveness of a behavioral medicine intervention in physical therapy on secondary psychological outcomes and health-related quality of life in exercise-based cardiac rehabilitation: a randomized, controlled trial. BMC Sports Sci Med Rehabil. 2023 Mar 24;15(1):42. doi: 10.1186/s13102-023-00647-x. PMID 36964593
- [Derived] Freene N, Borg S, McManus M, Mair T, Tan R, Davey R, Oberg B, Back M. Comparison of device-based physical activity and sedentary behaviour following percutaneous coronary intervention in a cohort from Sweden and Australia: a harmonised, exploratory study. BMC Sports Sci Med Rehabil. 2020 May 9;12:17. doi: 10.1186/s13102-020-00164-1. eCollection 2020. PMID 32419950
- [Derived] Borg S, Oberg B, Nilsson L, Soderlund A, Back M. The role of a behavioural medicine intervention in physiotherapy for the effects of rehabilitation outcomes in exercise-based cardiac rehabilitation (ECRA) - the study protocol of a randomised, controlled trial. BMC Cardiovasc Disord. 2017 May 25;17(1):134. doi: 10.1186/s12872-017-0557-7. PMID 28545400